CLINICAL TRIAL: NCT02490878
Title: Randomized Phase II Study: Corticosteroids + Bevacizumab vs. Corticosteroids + Placebo (BEST) for Radionecrosis After Radiosurgery for Brain Metastases
Brief Title: Corticosteroids + Bevacizumab vs. Corticosteroids + Placebo (BEST) for Radionecrosis After Radiosurgery for Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A221208; NCI-2015-01348 (Registry Identifier: NCI Clinical Trials Reporting Program); NCT02531659 (obsolete NCT alias)
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Results first posted 2021-08-06 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-02

CONDITIONS: Radionecrosis; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Bevacizumab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bevacizumab + corticosteroids (Experimental): The patient will receive bevacizumab 10 mg/kg IV given on days 1 and 15 of a 28 day cycle for 4 cycles. Once the patient has started the study treatment, the dose of corticosteroids will be tapered every 5 days (e.g., dexamethasone 2 mg or prednisone 15 mg per taper), as tolerated, under the management of the treating MD. If patients deteriorate while tapering, dexamethasone will be increased up to a maximum of 16 mg per day, as per treating MD, to manage symptoms.
  Patients who meet the criteria for clinical progression will be treated as per treating MD.
  Interventions: Drug: bevacizumab; Drug: corticosteroids
- placebo + corticosteroids (Experimental): The patient will receive placebo 0.9% NaCl volume equal to bevacizumab volume added to 100 mL bag of 0.9% NaCl delivered IV given on days 1 and 15 of a 28-day cycle for 4 cycles. Once the patient has started the study treatment, the dose of corticosteroids will be tapered every 5 days (e.g., dexamethasone 2 mg or prednisone 15 mg per taper), as tolerated, under the management of the treating MD. If patients deteriorate while tapering, dexamethasone will be increased up to a maximum of 16 mg per day, as per treating MD, to manage symptoms.
  Patients who meet the criteria for clinical progression will be allowed to receive bevacizumab according to the protocol.
  Interventions: Drug: corticosteroids; Other: placebo

INTERVENTIONS:
Drug: bevacizumab — IV
  Arms: bevacizumab + corticosteroids
Drug: corticosteroids — IV
Other: placebo — IV
  Arms: placebo + corticosteroids

SUMMARY:
This randomized phase II study aims to investigate whether the addition of bevacizumab to standard corticosteroid therapy results in greater improvement in symptoms and less treatment-induced symptoms compared with standard corticosteroid therapy for patients with symptomatic brain radionecrosis following radiosurgery. It is hypothesized that the addition of bevacizumab to standard care corticosteroids will reduce treatment-induced toxicities and improve neurologic impairments in patients with brain radionecrosis following radiosurgery for brain metastases.

DETAILED DESCRIPTION:
This is a randomized double-blinded phase II study of corticosteroids with bevacizumab vs. corticosteroids with placebo for brain radionecrosis following radiosurgery for brain metastases. This is a two-arm clinical trial with parallel group design for longitudinal quality of life endpoint. Patients will be stratified according to age (≤ 65 years vs. > 65 years), pathological confirmation of necrosis (yes vs. no), MDASI-BT mean global score (symptom + interference scores) ( < 4.0 vs. > 4.0) and prior whole brain radiotherapy (yes vs. no). The primary and secondary objectives are detailed below.

Primary Objective:

To investigate whether the addition of bevacizumab to standard corticosteroid therapy results in greater improvement in symptoms (clinical and patient-reported symptom improvement associated with radionecrosis and less radionecrosis treatment-induced symptoms) compared with standard corticosteroid therapy.

Secondary Objectives:

1. To evaluate the toxicity profile associated with bevacizumab and corticosteroid therapy.
2. To compare self-reported health related quality of life (HRQOL) using LASA, Dexamethasone Symptoms Questionnaire-Chronic (DSQ-C), and MDASI-BT symptom and interference score between treatment arms.
3. To compare intracranial progression-free survival and time to maximum radiographic response between treatment arms.
4. To compare the dose and duration of corticosteroids required between treatment arms and correlate steroid requirement with DSQ-C and MDASI-BT scores.

Patient event monitoring will occur every 2 months after treatment up to 6 months. Then event monitoring will occur up to one year.

ELIGIBILITY:
Pre-Registration Eligibility Criteria:

1. Patients who present with symptomatic brain radionecrosis after they have received radiosurgery for brain metastases from primary solid tumor including but not limited to lung, breast, colorectal cancer but excluding melanoma, choriocarcinoma, renal cell carcinoma or gliomas
2. Patients at institutions that elect to utilize central imaging review to confirm eligibility must be pre-registered prior to submission of these images; images should be submitted as soon as possible after the pre-registration magnetic resonance imaging (MRI) is obtained; turnaround time for this review will be =< 72 business hours after receipt of images by the Imaging and Radiation Oncology Core (IROC)
3. Patients at institutions that elect to confirm eligibility locally may be pre-registered at the same time as they are randomized

Registration/Randomization Eligibility Criteria:

1. A diagnosis of radionecrosis will be based on a clinical onset of symptoms and radiological findings of radionecrosis at 3-24 months following radiosurgery, with or without pathological confirmation.

   1.1 'Symptomatic' brain radionecrosis to at least one lesion following radiosurgery treatment for brain metastases where 'symptomatic' is defined as:

   1.1.1 New or increasing headache associated with mass effect, sensory or motor abnormality, cognitive changes, speech difficulty, balance or coordination difficulty, cranial nerve deficits

   1.1.2 Symptoms are persistent or worsening despite administration of at least dexamethasone 4 mg (or equivalent corticosteroid) daily for 1 week

   1.2 Clinical eligibility supported by central imaging real-time review. The presence of at least the following conventional MR image characteristic:

   1.2.1 Conventional MR - Lesion quotient of < 0.3, where lesion quotient is defined as the proportional value of the maximum axial cross-sectional area of the T2-weighted defined lesion over the maximum axial cross-sectional area of the contrast-enhancing lesion on the T1-weighted post-gadolinium sequence on a comparable axial slice. If the conventional MR findings are not seen, the following dynamic susceptibility-contrast (DSC) MR characteristics may be used to meet eligibility for this study.

   1.2.2 DSC MR - The cut-offs below will be based on GRE EPI DSC perfusion images, acquired without using a gadolinium pre-load:

   1.2.2.1 Relative cerebral blood volume (rCBV) <1.5 in the enhancing- lesion relative to normal-appearing white matter (NAWM)

   1.2.2.2. Percentage of signal recovery (PSR) > 76%, where PSR is determined by comparing the lower signal intensity during passage of the contrast bolus with the post-contrast signal intensity on the signal intensity-time curve

   1.2.3 Centers that standardly use PET or MRS to determine a diagnosis of radionecrosis are permitted to use these modalities to assist in their patient selection; however the criteria described for conventional MR and/or DSC should also be met for study eligibility. Both PET and MRS are not mandatory for study eligibility.
2. Prior to start of treatment

   2.1 Must have been taking a stable dose of corticosteroids for symptom management for at least 1 week before baseline MRI.

   2.2 No systemic therapy within 2 weeks prior to registration or plan for systemic therapy within the first 8 weeks after study registration. The protocol provides a list of 'approved systemic' therapies that are allowed for concurrent use with bevacizumab.

   2.3 No bevacizumab ≤ 3 months of study registration.

   2.4 Central imaging real-time review (72 hour turn around) to confirm eligibility.
3. Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown. Therefore, for women of childbearing potential only, a negative urine or serum pregnancy test done ≤ 14 days prior to registration and confirmation they are not nursing is required.
4. Age ≥ 18 years
5. Karnofsky Performance Status ≥ 60%
6. Required Initial Laboratory Values ≤14 days of registration:

   6.1 Absolute Neutrophil Count (ANC) ≥ 1,500/mm^3

   6.2 Platelet Count ≥ 100,000/mm3

   6.3 Hemoglobin ≥ 10 g/dL*

   6.3.1 allowing transfusion or other intervention to achieve this minimum hemoglobin

   6.4 BUN < 30 mg/dL

   6.5 Creatinine < 1.7 mg/dL

   6.6 Bilirubin ≤ 2.0 mg/dL

   6.7 ALT ≤ 3.0 x upper limits of normal (ULN)

   6.8 AST ≤ 3.0 x ULN

   6.9 INR <1.5 x ULN**

   6.9.1 unless patients are receiving anti-coagulation therapy. Patients receiving anti-coagulation therapy with an agent such warfarin or heparin are allowed to participate if INR ≤ 3.0.**

   6.10 UPC Ratio <0.5 or if ≥ 0.5

   6.10.1 24-hour urine protein must be <1000 mg
7. Able to participate in patient-report outcomes (MDASI-BT, DSQ-C, LASA) questionnaires.

   Assistance by research personnel is acceptable if participant has disabilities that make reading or writing difficult.
8. No evidence of recent hemorrhage at pre-registration MRI of the brain, however the following are permitted: presence of hemosiderin, resolving hemorrhagic changes related to surgery, and presence of punctate hemorrhage in the tumor.
9. No excess risk of bleeding (any of the following):

   9.1 Bleeding diathesis or coagulopathy

   9.2 Thrombocytopenia

   9.3 Major surgical procedure, open biopsy, or significant traumatic injury within the past 28 days or anticipation of need for major surgical procedure during the course of the study.

   9.4 Minor surgical procedures, stereotactic biopsy, fine needle aspiration, or core biopsy within the past 7 days.
10. No clinically significant cardiovascular disease.

    10.1 No uncontrolled hypertension (systolic blood pressure ≤ 160 mm Hg or diastolic ≤ 100 mm Hg). Patients with hypertension must be adequately controlled with appropriate anti-hypertensive therapy or diet.

    10.2 No history of arterial thrombotic events within the past 6 months, including:

    10.2.1 transient ischemic attack (TIA)

    10.2.2 cerebrovascular accident (CVA)

    10.2.3 peripheral arterial thrombus

    10.2.4 unstable angina or angina requiring surgical or medial intervention

    10.2.5 myocardial infarction (MI)

    10.2.6 significant peripheral artery disease (i.e., claudication on less than one block)

    10.2.7 significant vascular disease (i.e., aortic aneurysm, history of aortic dissection)

    10.3 Patients who have had a deep vein thrombosis or pulmonary embolus within the past 6 months are eligible if they are on stable therapeutic anticoagulation.

    10.4 No current New York Heart Association classification II, III, or IV congestive heart failure.
11. No history of bowel obstruction, abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within past 12 months.
12. No central lung metastases with excessive active bleeding.
13. No uncontrolled intercurrent illness including, but not limited to any of the following:

    ongoing or active infection requiring IV antibiotics, cardiac arrhythmia, or psychiatric illness and/or social situations that would limit compliance with study requirements.
14. No history of serious non-healing wound, ulcer, or bone fractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Chung, MD, Study Chair — M.D. Anderson Cancer Center
Locations (341):
- United States (332):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Mercy Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - William Beaumont Hospital-Grosse Point, Grosse Pointe, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Lymphoma Clinic of Michigan, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon and Rectal Association, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Saint Joseph Health System-Tawas City, Tawas City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Bhadresh Nayak MD PC-Warren, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Nevada Cancer Specialists-Saint Rose, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - Nevada Cancer Specialists?Oakey, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Nevada Cancer Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Specialists-Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - University of Rochester, Rochester, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physicians LLC-Samaritan North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates-Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates PA-Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Laurens, Clinton, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Ashland Memorial Medical Center, Ashland, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (9):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 patients underwent pre-screening. Only 19 underwent randomization.
Groups:
- Arm A: Bevacizumab: The patient will receive bevacizumab 10 mg/kg IV given on days 1 and 15 of a 28 day cycle for 4 cycles. Once the patient has started the study treatment, the dose of corticosteroids will be tapered every 5 days (e.g., dexamethasone 2 mg or prednisone 15 mg per taper), as tolerated, under the management of the treating MD. If patients deteriorate while tapering, dexamethasone will be increased up to a maximum of 16 mg per day, as per treating MD, to manage symptoms.
- Arm B: Placebo: The patient will receive placebo 0.9% NaCl volume equal to bevacizumab volume added to 100 mL bag of 0.9% NaCl delivered IV given on days 1 and 15 of a 28-day cycle for 4 cycles. Once the patient has started the study treatment, the dose of corticosteroids will be tapered every 5 days (e.g., dexamethasone 2 mg or prednisone 15 mg per taper), as tolerated, under the management of the treating MD. If patients deteriorate while tapering, dexamethasone will be increased up to a maximum of 16 mg per day, as per treating MD, to manage symptoms.
Period: Overall Study
Arm/Group | Arm A: Bevacizumab | Arm B: Placebo
Started | 10 | 9
Eligible Participants | 10 | 8
Completed | 10 | 6
Not Completed | 0 | 3
Not completed — deemed ineligible | 0 | 1
Not completed — progression prior to treatment | 0 | 1
Not completed — only submitted baseline QOL | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Bevacizumab | Arm B: Placebo | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Customized [Count of Participants; unit: Participants]
  Age group: <= 65 years | 7 | 5 | 12
  Age group: > 65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Prior whole brain radiotherapy [Count of Participants; unit: Participants]
  Yes | 5 | 1 | 6
  No | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in M. D. Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom Severity Score
Description: The MD Anderson Symptom Inventory for brain tumor (MDASI-BT) is a 28-item multi-symptom patient-reported outcome measure assessing the severity of symptoms experienced by cancer patients and the interference with daily living caused by these symptoms, with 9 items specific to brain tumors. Each item ranges from 0 (best condition) to 10 (worst condition). A subscale score (Symptom Severity) is the average of the subscale items with 0 being "not present" and 10 being "as bad as you can imagine.", given that a specified minimum numbers of items were completed. A negative change in score from baseline to given time point indicates a worsening score.
Time Frame: Baseline, 2, 4, 6 and 8 weeks
Population: All eligible patients that began protocol treatment and were assessed at baseline and at least one subsequent time within the first 8 weeks were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Bevacizumab | Arm B: Placebo
Number analyzed (Participants) | 10 | 6
score on a scale
  2 weeks | -0.8 (1.93) | 0.1 (1.24)
  4 weeks: number analyzed (Participants) | 8 | 4
  4 weeks | -0.5 (2.17) | -2.0 (2.53)
  6 weeks: number analyzed (Participants) | 8 | 3
  6 weeks | -0.5 (2.33) | -2.3 (2.86)
  8 weeks: number analyzed (Participants) | 7 | 2
  8 weeks | -0.6 (2.13) | -3.9 (2.83)

2. Secondary Outcome: Toxicity (CTCAE Version 4.0)
Description: Toxicity associated with bevacizumab and corticosteroids in patients with radionecrosis using CTCAE Version 4.0. The number of patients reporting a grade 3 or higher, 4 or higher, or 5 at least possibly related to treatment are included in this table.
Time Frame: Up to 1.5 years post-treatment
Population: All patients that began treatment are included in this endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Bevacizumab | Arm B: Placebo
Number analyzed (Participants) | 10 | 8
Participants
  Grade 3 or higher | 2 | 5
  Grade 4 or higher | 0 | 0
  Grade 5 | 0 | 0

3. Secondary Outcome: Quality of Life Measure Using the Single Item Linear Analogue Scale (LASA)
Description: The Linear Analogue Scale used is a 5-question survey. Patients are asked to score the following questions on a 1(as bad as it can be) -10 (as good as it can be) scale: 1) your overall quality of life, 2) your overall (intellectual) well being, 3) your overall physical well being, 4) your overall emotional well being, and 5) your overall spiritual well being. The change in score was computed from baseline to 1.5 years post-treatment. A negative difference is thought of as a worsening score from baseline.
Time Frame: Up to 1.5 years post-treatment
Population: All patients that completed the LASA at baseline and at 1.5 years after treatment were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Bevacizumab | Arm B: Placebo
Number analyzed (Participants) | 8 | 5
score on a scale
  LASA Overall Quality of Life | -1.0 (3.07) | 0.0 (2.55)
  LASA Mental well being | -1.5 (3.12) | 0.0 (1.73)
  LASA Physical well being | -1.1 (3.4) | 0.4 (1.14)
  LASA Emotional well being | -1.0 (2.45) | 1.8 (3.03)
  LASA Spiritual well being | -1.1 (2.42) | 0.8 (2.17)

4. Secondary Outcome: Quality of Life Measure Using the Dexamethasone Symptoms Questionnaire - Chronic (DSQ-C)
Description: The DSQ-C was developed for use in the brain tumor patient population. It consists of 18 questions rated on a 4-point scale (1 to 4, with 4 indicating a worse symptom) to indicate the presence and severity of symptoms. For each patient, the sum across all 18 questions were computed(18-72, with 18 being a score of 1 for each of the 18 questions and 72 being a score of 4 for each of the questions, refering to the previous sentence, a score of 18(a score of 1, 18 times) indicates the best possible score. A score of 72(a score of 4, 18 times) indicates the worst possible. The mean for total score across each week (weeks 2, 4, 6, 8) is reported.
Time Frame: Baseline and weeks 2, 4, 6, 8 of treatment
Population: All patients that received protocol treatment and completed the survey at baseline were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Bevacizumab | Arm B: Placebo
Number analyzed (Participants) | 10 | 7
score on a scale
  Baseline | 1.0 (0.15) | 1.2 (0.33)
  Week 2: number analyzed (Participants) | 10 | 6
  Week 2 | 1.0 (0.14) | 1.2 (0.23)
  Week 4: number analyzed (Participants) | 8 | 4
  Week 4 | 1.0 (0.14) | 1.0 (0.14)
  Week 6: number analyzed (Participants) | 8 | 3
  Week 6 | 1.0 (0.07) | 1.0 (0.07)
  Week 8: number analyzed (Participants) | 7 | 2
  Week 8 | 1.0 (0.15) | 1.0 (0.16)

5. Secondary Outcome: Quality of Life Measure Using the The M. D. Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) Score.
Description: The MDASI-BT was developed and validated for use in the brain tumor patient population, including those with brain metastases and typically requires less than 4 minutes to complete. It consists of 23 symptoms rated on a 0 to 10 numerical rating scale (NRS) to indicate the presence and severity of the symptom, with 0 being "not present" and 10 being "as bad as you can imagine." MDASI-BT Symptom Scoring: A global symptom score for the MDASI symptom severity scale is obtained by taking the average of the 23 items together. This puts the score on a 0-10 scalenumerical rating scale (NRS) to indicate the presence and severity of the symptom, with 0 being "not present" and 10 being "as bad as you can imagine." The mean global symptom at baseline and at weeks 2, 4, 6, 8 were used in this analysis.
Time Frame: Up to 1.5 years post-treatment
Population: All patients that began protocol treatment and completed the survey at study entry or within 8 weeks were included in this analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Bevacizumab | Arm B: Placebo
Number analyzed (Participants) | 10 | 6
score on a scale
  Baseline | 4.0 (1.51) | 5.3 (2.27)
  Week 2 | 2.9 (2.39) | 6.1 (0.88)
  Week 4 | 3.9 (2.75) | 4.8 (1.73)
  Week 6 | 3.9 (2.21) | 4.9 (3.29)
  Week 8 | 4.0 (2.44) | 4.3 (3.06)

6. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the time from start of treatment to the earliest of the date patient stops placebo or bevacizumab for either alternative therapy or crossover to bevacizumab (if initially on placebo). Result will be summarized by Kaplan-Meier method.
Time Frame: Up to 16 weeks
Population: All patients that registered were included in this analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A: Bevacizumab | Arm B: Placebo
Number analyzed (Participants) | 10 | 9
days | NA [NA to NA] — Too few events have been reported to obtain a median or estimate a 95% Confidence Interval | NA [103.0 to NA] — Too few events have been reported to obtain a median or estimate an upper level 95% Confidence Interval

7. Secondary Outcome: Time to Maximum Radiographic Response
Description: Time from start of treatment to maximum radiographic response
Time Frame: Up to 16 weeks
Population: Due to early trial termination data was not collected and could not be analyzed.
Arm/Group | Arm A: Bevacizumab | Arm B: Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time to Stopping Corticosteroids
Description: Time to stopping corticosteroids is defined as the time from start of protocol treatment to the last day corticosteroids were given. Time to stopping corticosteroid will be summarized by Kaplan-Meier curve with log-rank tests conducted to investigate differences between treatment arms.
Time Frame: Up to 16 weeks
Population: All patients that registered for treatment were included in this analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A: Bevacizumab | Arm B: Placebo
Number analyzed (Participants) | 10 | 9
days | 113 [50 to 141] | 102 [29 to 252]

ADVERSE EVENTS:
Time Frame: Adverse events were collected on days 1 and 15 during 4 cycles of treatment. Each cycle was 28 days.
Arm/Group | Arm A: Bevacizumab | Arm B: Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/8
Serious Adverse Events (participants affected / at risk) | 3/10 | 6/8
Other Adverse Events (participants affected / at risk) | 10/10 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Bevacizumab (N=10) | Arm B: Placebo (N=8)
Fever (General disorders) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (3)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Bevacizumab (N=10) | Arm B: Placebo (N=8)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (6)
Cushingoid (Endocrine disorders) | 1 (3) | 0 (0)
Blurred vision (Eye disorders) | 1 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (4) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (4) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (12) | 4 (12)
Gait disturbance (General disorders) | 2 (2) | 1 (2)
Localized edema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (3) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 1 (8)
Weight gain (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 1 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2)
Facial nerve disorder (Nervous system disorders) | 1 (2) | 0 (0)
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 1 (4)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 7 (43) | 7 (19)
Hypotension (Vascular disorders) | 1 (2) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT02490878/Prot_SAP_ICF_000.pdf